CLINICAL TRIAL: NCT00663520
Title: Elucidating the Role of Microvascular Dysfunction in Heart Disease in Women
Acronym: MVD
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Elizabeth Cannar, Diana Rinkevich, MD, Oregon Health and Science University
Other Study IDs: Study #3631
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Microvascular Dysfunction
Keywords: Cardiac disease; vascular dysfunction; women; chest pain; echocardiography
MeSH Terms: conditions — Heart Diseases; Chest Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Women with chest pain and "Clean" heart vessels
- 2: Healthy volunteers

SUMMARY:
The purpose of this study is to determine if women with chest pain and "clean" heart blood vessels have impaired blood flow to the heart due to problems with the small blood vessels that provide blood and oxygen to the heart. Impairment in the small blood vessels will be tested using ultrasound pictures of the heart, called myocardial contrast echocardiography. Since these small blood vessels are not seen in a coronary angiogram, which is an x-ray of the heart vessels using a dye containing iodine injected in the heart vessels, the problem may remain undiagnosed in women until the heart muscle becomes severely damaged.

A second purpose is to identify if there is a common trait in the population of women with this tiny blood vessel dysfunction, which will be investigated by checking blood levels of certain chemical and hormones related to heart disease. Finally, we would like to investigate the relationship between depression and stress, and heart disease. We will do this by measuring cortisol (a hormone that serves as a measure of stress) and administering questionnaires that help to identify depression and stress.

ELIGIBILITY:
Inclusion Criteria:

* Women 45 to 75 years of age

Exclusion Criteria:

* Pregnancy
* Allergy to any component of the drugs: Definity®. Dipyridamole Aminophyllin or Iodine.
* Known coronary heart disease, significant valvular disease (valvular stenosis or insufficiency greater than moderate) left ventricular systolic dysfunction, congenital heart disease or cardiac shunt, pulmonary hypertension, moderate or severe asthma.
* Inability to reach the patient by mail, fax, e-mail or phone
* Active infection
* Malignancy
* Uncontrolled hypertension
* Smoking
* Severe asthma
* Kidney disease

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifty non-smoking women, between 45 and 75 years of age, with chest pain will be referred to this study by clinicians at OHSU. The control group will be fifty non-smoking women with no cardiac symptoms, matched with the study group by age and risk factors. Flyers and other advertisements may be used to recruit both the study group and the control group. Criteria for exclusion from the study are pregnancy, allergy to any component in the drugs used in the study, severe asthma, known disease of the heart vessels or heart valves, active infection, cancer, uncontrolled hypertension, kidney disease and current smoking status.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Elucidating the Role of Microvascular Dysfunction in Heart Disease in Women | 2008-2014
  Data collection

CONTACTS AND LOCATIONS:
Overall Officials: Diana Rinkevich, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
No Plan to share data.